CLINICAL TRIAL: NCT06128096
Title: The Effect of SGLT-2 Inhibitors on Epicardial Adipose Tissue and Cardiac Function in T2DM Patients With CAD (EpiCAD)
Acronym: EpiCAD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Clinical Research Centre, Malaysia (Other)
Collaborators: University of Malaya (Other); Ministry of Health, Malaysia (Other Government)
Responsible Party: Principal Investigator, Wan Ahmad Syazani bin Mohamed, Principal Investigator, Clinical Research Centre, Malaysia
Other Study IDs: NMRR ID-22-02966-ENM
Record Dates: First submitted 2023-11-07; First posted 2023-11-13 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; SGLT-2 Inhibitor; Antidabetic Agent; Cardiac Function; Epicardial Adipose Tissue
MeSH Terms: conditions — Coronary Artery Disease | interventions — dapagliflozin; empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For DNA extraction and RT-PCR (Pharmacogenomic) - Only for 6 months follow up to evaluate pharmacogenomic of treated patients and controls
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- SGLT-2 inhibitor group: Patients will be given a recommended dose of SGLT-2 inhibitor by cardiologist in a form of tablets based on clinical indication. The SGLT-2 inhibitor includes :
  1. Tab Empagliflozin 10mg OD
  2. Tab Dapagliflozin 10mg OD
  After administration of SGLT-2 inhibitor, the cardiac function and epicardial adipose tissue thickness will be measured (baseline and 6 month) post intervention
  Interventions: Drug: Sodium Glucose Co-transporter 2 (SGLT2) Inhibitor
- Control group: Patient will not be given SGLT-2 inhibitor and continue SOC up to 6 months. The cardiac function and epicardial adipose tissue thickness will be measured (baseline and 6 month) post intervention

INTERVENTIONS:
Drug: Sodium Glucose Co-transporter 2 (SGLT2) Inhibitor — Patients (180 diabetic patients with CAD that are using SGLT-2 inhibitors and 180 diabetic patients with CAD that are not using SGLT-2 inhibitors) who fulfil the inclusion and exclusion criteria will be recruited from the following sources:
  UMMC Cardiology and Diabetes out-patient clinics UMMC Cardiology and Endocrinology in-patients (wards)
  During the recruitment, patients will do baseline echocardiography in which includes epicardial adipose tissue and cardiac function. The same procedure will be repeated 6 months post intervention.
  Other Names: Forxiga (Dapagliflozin); Jardiance (Empagliflozin)
  Groups: SGLT-2 inhibitor group

SUMMARY:
Sodium-glucose contrasporter-2 (SGLT-2) inhibitors make up an antidiabetic medication that promotes glycosuria. They are known to have an indirect reduction in cardiovascular complications, based on a series of in-depth studies. However, the effect of SGLT-2 inhibitors towards the thickness of epicardial adipose tissue and cardiac function in type 2 diabetes mellitus (T2DM) with coronary artery disease (CAD) patients in Malaysia has not yet been fully explored. Therefore, this study aims to determine the effects in epicardial adipose tissue thickness and its cardiac function in T2DM patients with CAD after the initiation of SGLT-2 inhibitors.

DETAILED DESCRIPTION:
Type 2 diabetes mellitus (T2DM) is a chronic metabolic disorder affecting at least 90% of the population with diabetes globally (Bhupathiraju & Hu, 2016). T2DM is a disorder characterized insulin resistance, insufficient insulin production, and eventual pancreatic beta-cell failure (Cantley & Ashcroft, 2015).The global prevalence of T2DM has been increasing steadily, with an estimate of 463 million individuals suffering from T2DM in 2019 and the number is projected to increase by 15.7% in 2030 (Saeedi et al., 2019). T2DM is also increasing at an alarming rate in Malaysia and as of 2019 (Akhtar et al., 2022), approximately 3.5 million (17.5%) Malaysians were diagnosed with T2DM, which doubled in number since 1996 (8.3%) (Zhu et al., 2019).

Evidently, T2DM patients are predisposed to various forms of both short and long-term complication, with cardiovascular disease (CVD) being the main cause of death among T2DM patients (Raghavan et al., 2019), T2DM has been shown to decrease life expectancy by 10 years with CVD responsible for half of the mortality (Einarson et al., 2018). Although a close link between T2DM and CVD is established, the etiology is complex and remains a significant research topic. Obesity, traditionally defined as excess body weight and adiposity, is closely linked to the pathogenesis of T2DM. Obesity associated with T2DM is linked with a cluster of metabolic and biochemical abnormalities with insulin resistance central in promoting these disturbances. It could manifest itself in various pathophysiological states which includes hyperglycemia, atherogenic dyslipidemia, inflammation, and endothelial dysfunction (Galicia-Garcia et al., 2020). These pathological states have been shown to exacerbate the progression of CVD; and according to a global systematic review, patients with T2DM had a 10% greater risk of coronary artery disease (CAD), approximately 50% higher risk of developing myocardial infarction (MI) and stroke, and a staggering 112% increased risk for heart failure (Einarson et al., 2018).

The discovery of new pharmacotherapy to reduce complications associated with T2DM has brought global attention to sodium-glucose co-transporter 2 (SGLT-2) inhibitors, a relatively new anti-diabetic medication. SGLT-2 inhibitor exerts its hypoglycemic action by primarily blocking glucose reabsorption in the proximal convoluted tubule of the kidney which subsequently leads to glycosuria. This, in turn, promotes the utilization of lipids for energy production in response to high glucose lost resembling prolonged fasting state(Ferrannini et al., 2016; Yokono et al., 2014; Zaccardi et al., 2016). Due to these metabolic changes, SGLT-2 inhibitors reportedly induce weight loss due to its ability to reduce visceral and subcutaneous adipose tissues accumulation (Bramante et al., 2020; Pereira & Eriksson, 2019). Evidently, a clinical trial conducted by Zinman et al. (2016) reported remarkable reduction of cardiovascular-related mortality, and decreased risk of hospitalization and re-hospitalization for heart failure in T2DM patients receiving SGLT-2 inhibitors. In addition, one meta-analysis conducted by Zheng et al. (2018) also demonstrated that SGLT-2 inhibitors are able to reduce all-cause mortality in T2DM patients with CAD. Thus, emerging evidence suggested that SGLT-2 inhibitors are capable of decreasing the occurrence of cardiovascular events in T2DM patients, and closely linked to their ability to reduce fat content (Scheen, 2014).

As the indirect target of SGLT-2 inhibitors is towards reduction of adiposity, adipose tissue measurements were also shown to be an important indicator of SGLT-2 inhibitors effectiveness. According to Singh et al. (2007), visceral adipose tissue (VAT) which surrounds the internal organs of body cavities, could predict an undesirable metabolic and cardiovascular risk stratification. For this reason, epicardial adipose tissue (EAT), a type of visceral fat surrounding the heart supplied by major branches of coronary vessels, is increasingly studied to be the measuring point for the efficacy of SGLT-2 inhibitors (Sato et al., 2018; Yagi et al., 2017).

EAT originates from splanchnopleuric mesoderm, in which embryonically similar to intraabdominal adipose tissue and actively produces numerous cytokines that are essential for metabolic homeostasis (Muñoz et al., 2014). Physiologically, normal EAT distribution is required to provide a protective physiological role to the heart (Iacobellis et al., 2008). Normal EAT thickness is reported to be between 4.5mm- 7.0mm (Iacobellis et al., 2008). Physiologically, normal EAT thickness provides protective metabolic and thermogenic function towards both myocardium and coronary arteries (Wu et al., 2017; Iacobellis & Willens, 2009). EAT also produces adipokines, a signaling protein that regulates lipid and glucose-insulin metabolism in the heart (Talman et al., 2014; Wu et al., 2017). However, excessive EAT depot has been hypothesized to be involved in the pathogenesis and the progression of coronary artery disease, with the release of inflammatory mediators which prompt the atherosclerotic process through several paracrine mechanisms (Alexopoulos et al., 2010). Apart from metabolic disorders, there are various determinants that can contribute to EAT thickness, including age, gender, race and ethnicities (Lima-Martínez et al., 2014; Verma et al., 2017). Given that the estimation of cardiovascular risk is significantly relevant with EAT as compared to other visceral fat, the SGLT-2 anti-obesity effect on EAT accumulation may serve as a significant cardiovascular predictor in T2DM patients (Sato et al., 2018; Yagi et al., 2017).Evidently, due its significant metabolic effect, SGLT-2 inhibitors have also been shown to reduce the amount of visceral adipose tissue by caloric elimination and thereby reducing EAT in multiple pilot studies (Fukuda et al. 2017; Braha et al. 2019; Yagi et al. 2017).

Given its anatomical proximity to the heart, EAT is now proposed to be more relevant cardiovascular risk estimation than other visceral fat depot, with multiple emerging studies have demonstrated that EAT is associated with increased coronary artery calcification (Mancio et al., 2017). Parallel to this, our preliminary study from UMMC cardiology patients indicated that patients with CAD have significantly thicker EAT, and positively correlated with BMI. Given the emerging role of SGLT-2 inhibitors as treatment for obesity, its effect in reducing visceral fat, particularly on EAT, is increasingly studied. But its role specifically in T2DM and how it can be developed as a therapeutic target to reduce CVD risk among our high-risk population in our local clinical setting is less understood. Therefore, the aim of this study is to investigate the effect of SGLT-2 inhibitors on EAT thickness, metabolic outcomes and subsequently cardiac function in T2DM patients.

More significantly, currently, there are no existing studies which report the EAT distribution with other cardiac function parameters among Malaysian and its clinical implication in the local clinical setting. Our preliminary study from UMMC cardiology patients also indicated that Malay male have significantly thicker EAT compared to other ethnicities. Indeed, measures of total body fat and depot-specific adiposity reveal distinct ethnic patterns, which may portend different health implications (Staiano et al., 2013), particularly among multi-ethnics Malaysians. In addition, the associations between EAT thickness and cardiac function among ethnic-diverse Malaysian T2DM patients receiving SGLT-2 inhibitors are yet to be explored. Thus, the current study hopes to conclude the link of evidences between EAT and cardiac function in T2DM patient with CAD that were receiving SGLT-2 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Malaysian patients aged 18 years old and above.
* Diagnosed with type 2 diabetes mellitus and not any other types of diabetes.
* Established diagnosis of coronary artery disease. * (see definition below)
* Glomerular filtration rate (GFR) >30ml/min/1.73m2
* Women that are not pregnant or breastfeeding during recruitment.
* Initiated with SGLT-2 inhibitors for not more than 3 months before recruitment or initiating SGLT-2 at the time of recruitment.

Exclusion Criteria:

* Patients that are contraindicated to SGLT-2 inhibitors
* Other types of diabetes aside from type 2 diabetes mellitus
* Initiated with SGLT-2 inhibitors for more than 3 months
* History of diabetes ketoacidosis
* History of repeated urinary infections or urogenital infections developed during the study
* Glomerular filtration rate (GFR) < 30ml/min/1.73m2 (Stage 4 and Stage 5 CKD)
* Other side effects that required discontinuation of treatment with SGLTs
* Patients with poor quality of echocardiogram image
* Patients with incomplete data of metabolic syndrome components.
* Patients who are not compliant
* Patient's refusal to take part in the study
* Any clinically significant findings or unstable condition during the screening, medical history, or physical examination that, in the investigator's opinion, would compromise participation in this study. This could include patients with poorly controlled hypertension, asthma, diabetes, or other life-threatening conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (180 T2DM patients that are using SGLT-2 inhibitors and 180 T2DM patients that are not using SGLT-2 inhibitors) who fulfil the inclusion and exclusion criteria will be recruited from the following sources:
  1. UMMC Cardiology and Diabetes out-patient clinics
  2. UMMC Cardiology and Endocrinology in-patients (wards)
  All recruited patients will have echocardiogram done during the day of recruitment. A repeated echocardiogram will be carried out at 6-month post recruitment.
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Left Ventricular Ejection Fraction | 6 months
  LVEF in %
Left Ventricular Mass Index | 6 months
  LVMI in gram
Left Ventricular Filling Pressure Ratio | 6 months
  E/e in ratio
Left Ventricular End Diastolic Diameter | 6 months
  LVEDD in centimeter
Left Ventricular End Systolic Diameter | 6 months
  LVESD in centimeter
Left Ventricular End Diastolic Volume | 6 months
  LVEDV in mililiter
Left Ventricular End Systolic Volume | 6 months
  LVESV in mililiter
Epicardial Adipose Tissue | 6 months
  Thickness of epicardial adipose tissue in milimeter

CONTACTS AND LOCATIONS:
Overall Officials: Wan Ahmad Syazani Mohamed, Principal Investigator — Institute For Medical Research (IMR), Malaysia
Locations (1):
- Institute for Clinical Research, National Institutes of Health, Malaysia, Shah Alam, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
Protocol can be shared with other researchers